CLINICAL TRIAL: NCT03302806
Title: Observational Study to Assess Effect and Safety of High Dose of Biotin (Qizenday®) in Progressive Multiple Sclerosis
Brief Title: Study to Assess Effect and Safety of High Dose of Biotin (Qizenday®) in Progressive Multiple Sclerosis
Acronym: BIOSEP
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0232
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Progressive Multiple Sclerosis
Keywords: disability; EDSS
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non interventional Study

SUMMARY:
The purpose of this observational study is to collect efficacy and safety data in real life condition within the first year of treatment in patients with progressive multiple receiving a daily dose of biotine of 300 mg.

ELIGIBILITY:
Inclusion Criteria:

* Progressive multiple sclerosis patients with an EDSS score ≤ 7 who have been prescribed high dose of biotin (temporary use administration) at Nantes university hospital (France)

Exclusion Criteria:

* Patient with remittent recurrent multiple sclerosis
* Pregnant women or women contemplating pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with progressive multiple receiving a daily dose of biotine of 300 mg
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Evolution of post-treatment disability | 12 months
  Change in Expanded Disability Status Scale (EDSS) progression from pretreatment period

SECONDARY OUTCOMES:
CGI-t scale | after 6 months and 12 months
  Change in Clinical global impression of improvement from both physician and patient assessments
Functional disability : Multiple sclerosis Functional composite | 12 months
  Composite score : Change in test measuring the patient's walking speed over a distance of 25 feet(TW25), Symbol Digit Modalities Test (SDMT), 9-Hole Peg Test Scores (9HPT) from baseline
Ambulation | 12 months
  Change in MSWS-12 score from baseline
Quality of life | 12 months
  Composite score : Change in EQ5D, MusiQuol, TLS coping 10 score from baseline
adverse effect (adverse drug reaction) | 12 months
  number of AE

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No